CLINICAL TRIAL: NCT00049036
Title: A Randomized Phase II Trial of EPOCH Given Either Concurrently or Sequentially With Rituximab in Patients With Intermediate- or High-Grade HIV-Associated B-cell Non-Hodgkin's Lymphoma
Brief Title: Combination Chemotherapy and Rituximab in Treating Patients With HIV-Associated Stage I, Stage II, Stage III, or Stage IV Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02926; NCI-2012-02926 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ECOG-AMC34; CDR0000257660; AMC-034 (Other: AIDS - Associated Malignancies Clinical Trials Consortium); AMC-034 (Other: CTEP); U01CA070019 (NIH)
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Results first posted 2011-06-22 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2012-12

CONDITIONS: AIDS-related Diffuse Large Cell Lymphoma; AIDS-related Immunoblastic Large Cell Lymphoma; AIDS-related Peripheral/Systemic Lymphoma; AIDS-related Small Noncleaved Cell Lymphoma
MeSH Terms: interventions — Rituximab; Etoposide; Doxorubicin; Vincristine; Prednisone; Cyclophosphamide

ARMS (2):
- Arm I (Experimental): Patients receive rituximab intravenously (IV) over 2-4 hours prior to each course of chemotherapy. Treatment repeats every 3 weeks for 4-6 courses. Patients who achieve a complete response after 4 courses of chemotherapy and rituximab receive additional rituximab alone weekly for 2 weeks.
  Interventions: Biological: rituximab; Drug: etoposide; Drug: doxorubicin hydrochloride; Drug: vincristine sulfate; Drug: prednisone; Drug: cyclophosphamide; Other: laboratory biomarker analysis
- Arm II (Experimental): Patients do not receive rituximab concurrently with chemotherapy. Beginning 4 weeks after completion of chemotherapy, patients receive rituximab IV over 2-4 hours weekly for 6 weeks.
  Interventions: Biological: rituximab; Drug: etoposide; Drug: doxorubicin hydrochloride; Drug: vincristine sulfate; Drug: prednisone; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: vincristine sulfate — Given IV
  Other Names: leurocristine sulfate; VCR; Vincasar PFS
Drug: prednisone — Given orally
  Other Names: DeCortin; Deltra
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
  Arms: Arm I
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial is studying how well giving combination chemotherapy together with rituximab works in treating patients with HIV-associated stage I, stage II, stage III, or stage IV non-Hodgkin's lymphoma. Drugs used in chemotherapy work in different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Combining chemotherapy with monoclonal antibody therapy may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the complete response rate after treatment with EPOCH given either concurrently or sequentially with rituximab.

SECONDARY OBJECTIVES:

I. To evaluate the toxicity of EPOCH given either concurrently or sequentially with rituximab.

II. To evaluate the effect of EPOCH given either concurrently or sequentially with rituximab on immune function (CD4, CD8 lymphocyte count) after two cycles of EPOCH, and 1 month, 3 months, 6 months, and 12 months after the completion of EPOCH.

III. To evaluate the effect of EPOCH given either concurrently or sequentially with rituximab on HIV and EBV viral load after two cycles of EPOCH, and 1 month, 3 months, 6 months, and 12 months after the completion of EPOCH.

IV. To evaluate the relationship between EBV viral load and EBV CD8 cytotoxic T cells in the peripheral blood and the presence of EBV in lymphoma tumor cells.

V. To determine whether rituximab or the concurrent use of antiretroviral therapy significantly alters the steady state concentration of etoposide, doxorubicin, or vincristine during the first cycle of therapy.

VI. To determine whether steady state concentration of etoposide or doxorubicin correlate with nadir neutrophil and platelet count during the first cycle of therapy.

VII. To determine time to progression and overall survival in patients treated with EPOCH given either concurrently or sequentially with rituximab.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to CD4 count (less than 100/mm^3 vs at least 100/mm^3), age-adjusted International Prognostic Index adverse risk factors (0 or 1 vs 2 or 3), and concurrent antiretroviral therapy (yes vs no). Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive rituximab intravenously (IV) over 2-4 hours prior to each course of chemotherapy. Treatment repeats every 3 weeks for 4-6 courses. Patients who achieve a complete response after 4 courses of chemotherapy and rituximab receive additional rituximab alone weekly for 2 weeks.

ARM II: Patients do not receive rituximab concurrently with chemotherapy. Beginning 4 weeks after completion of chemotherapy, patients receive rituximab IV over 2-4 hours weekly for 6 weeks.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated histologically or cytologically documented B-cell non-Hodgkin's lymphoma; the following histologies are eligible: diffuse large B-cell lymphoma, high-grade large cell immunoblastic lymphoma, anaplastic large cell lymphoma, Burkitt's lymphoma, high-grade B-cell lymphoma, Burkitt-like (small non-cleaved lymphoma)
* Tumors must be CD20 positive
* Documented HIV infection: documentation may be serologic (ELISA, western blot), culture, or quantitative PCR or bDNA assays
* Evaluable or measurable disease
* Stage I and IE or Stage II-IV disease patients
* ANC >= 1000 cells/mm^3
* Platelet count >= 75,000/mm^3 unless cytopenias are secondary to lymphoma
* All patients must be off colony stimulating factor therapy at least 24 hours prior to chemotherapy
* Transaminase =< 5 times the upper limit of normal unless secondary to hepatic infiltration with lymphoma or isolated hyperbilirubinemia associated with the use of indinavir or other antiretrovirals
* Total Bilirubin < 2.0 unless secondary to hepatic infiltration with lymphoma or isolated hyperbilirubinemia associated with the use of indinavir or other antiretrovirals; for bilirubin > 3.0 due to hepatic involvement the initial dose of doxorubicin will be decreased by 50% and the initial dose of vincristine will be omitted
* Creatinine < 2.0 unless due to lymphoma
* KPS >= 50 (ECOG PS 0, 1, or 2)
* Able to give consent
* Female patients must have a negative pregnancy test within 72 hours of entering into the study; males and females must agree to use adequate birth control if conception is possible during the study; women must avoid pregnancy and men avoid fathering children while in the study
* Patients already receiving erythropoeitin or G-CSF are eligible
* Patients must have a left ventricular ejection fraction that is at or above the lower institutional limits of normal, as assessed by nuclear scan or echocardiogram obtained within 12 weeks of registration
* Lymphomatous meningitis (patients with a positive CSF cytology are eligible)

Exclusion Criteria:

* Previous chemotherapy or radiotherapy for this lymphoma
* Primary Central Nervous System Lymphoma (parenchymal brain or spinal cord tumor)
* Acute active HIV-associated opportunistic infection requiring antibiotic treatment; patients with mycobacterium avium are not excluded; chronic therapy with potentially myelosuppressive agents is allowed provided that entry hematologic criteria are met
* Concurrent malignancy (excluding in situ cervical cancer, or non-metastatic non-melanomatous skin cancer, or Kaposi's sarcoma not requiring systemic chemotherapy)
* Previous therapy with rituximab within 12 months; patients treated with rituximab more than 12 months earlier are eligible only if it was given for indications other than the treatment of intermediate- or high-grade lymphoma (eg, low-grade lymphoma or ITP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2003-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Sparano, Principal Investigator — AIDS Associated Malignancies Clinical Trials Consortium
Locations (1):
- AIDS - Associated Malignancies Clinical Trials Consortium, Rockville, Maryland, United States

REFERENCES:
- [Derived] Sparano JA, Lee JY, Kaplan LD, Ramos JC, Ambinder RF, Wachsman W, Aboulafia D, Noy A, Henry DH, Ratner L, Cesarman E, Chadburn A, Mitsuyasu R. Response-adapted therapy with infusional EPOCH chemotherapy plus rituximab in HIV-associated, B-cell non-Hodgkin's lymphoma. Haematologica. 2021 Mar 1;106(3):730-735. doi: 10.3324/haematol.2019.243386. PMID 32107337
- [Derived] Sparano JA, Lee JY, Kaplan LD, Levine AM, Ramos JC, Ambinder RF, Wachsman W, Aboulafia D, Noy A, Henry DH, Von Roenn J, Dezube BJ, Remick SC, Shah MH, Leichman L, Ratner L, Cesarman E, Chadburn A, Mitsuyasu R; AIDS Malignancy Consortium. Rituximab plus concurrent infusional EPOCH chemotherapy is highly effective in HIV-associated B-cell non-Hodgkin lymphoma. Blood. 2010 Apr 15;115(15):3008-16. doi: 10.1182/blood-2009-08-231613. Epub 2009 Dec 18. PMID 20023215

RESULTS

PARTICIPANT FLOW:
Groups:
- EPOCH + Concurrent Rituximab: Patients receive rituximab IV over 2-4 hours prior to each course of chemotherapy. Treatment repeats every 3 weeks for 4-6 courses. Patients who achieve a complete response after 4 courses of chemotherapy and rituximab receive additional rituximab alone weekly for 2 weeks.
- EPOCH Followed by Rituximab: Patients do not receive rituximab concurrently with chemotherapy. Beginning 4 weeks after completion of chemotherapy, patients receive rituximab IV over 2-4 hours weekly for 6 weeks.
Period: Overall Study
Arm/Group | EPOCH + Concurrent Rituximab | EPOCH Followed by Rituximab
Started | 51 | 55
Completed | 51 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EPOCH + Concurrent Rituximab | EPOCH Followed by Rituximab | Total
Number analyzed (Participants) | 51 | 55 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 54 | 105
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (8.4) | 42.6 (9.4) | 42.6 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 43 | 48 | 91
Region of Enrollment [Number; unit: participants]
  United States | 51 | 55 | 106

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Proportion as Measured by Tumor Response After Completion of Study Treatment
Description: Complete response defined by the International Response Criteria for Non-Hodgkin's Lymphoma
Time Frame: 60 days
Population: ITT
Measure: Number; unit: proportion
Arm/Group | EPOCH + Concurrent Rituximab | EPOCH Followed by Rituximab
Number analyzed (Participants) | 51 | 55
proportion | 0.69 | 0.53

ADVERSE EVENTS:
Arm/Group | EPOCH + Concurrent Rituximab | EPOCH Followed by Rituximab
Serious Adverse Events (participants affected / at risk) | 28/51 | 27/55
Other Adverse Events (participants affected / at risk) | 50/51 | 51/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EPOCH + Concurrent Rituximab (N=51) | EPOCH Followed by Rituximab (N=55)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Anorexia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Autoimmune disorder (Immune system disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Bone infection (Infections and infestations) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1) | 3 (3)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (6) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Confusion (Nervous system disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Dehydration (General disorders) | 3 (10) | 2 (3)
Depressed level of consciousness (Nervous system disorders) | 1 (8) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 5 (5)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (9) | 0 (0)
ENT exam abnormal (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (8) | 7 (8)
Fever (General disorders) | 4 (12) | 5 (7)
Flu-like symptoms (Infections and infestations) | 1 (2) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 2 (2)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (6) | 1 (6)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemorrhage (Blood and lymphatic system disorders) | 2 (7) | 0 (0)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 3 (3) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 10 (20) | 6 (8)
Infectious meningitis (Infections and infestations) | 1 (1) | 0 (0)
Injection site reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 4 (12) | 6 (9)
Lymphatic disorder (General disorders) | 1 (2) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Multi-organ failure (General disorders) | 1 (9) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (8) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (6)
Neurological disorder (Nervous system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 9 (15) | 9 (10)
Pain (General disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Platelet count decreases (Blood and lymphatic system disorders) | 2 (7) | 2 (4)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (2) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (6) | 0 (0)
Seizure (Nervous system disorders) | 2 (9) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 1 (3) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (4)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EPOCH + Concurrent Rituximab (N=51) | EPOCH Followed by Rituximab (N=55)
Abdominal pain (Gastrointestinal disorders) | 14 (25) | 18 (40)
Alanine aminotransferase increases (Metabolism and nutrition disorders) | 13 (30) | 19 (62)
Alkaline phosphatase increases (Metabolism and nutrition disorders) | 11 (29) | 17 (43)
Allergic rhinitis (Immune system disorders) | 6 (19) | 5 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 16 (46) | 16 (39)
Anorexia (Gastrointestinal disorders) | 10 (24) | 10 (14)
Anxiety (Nervous system disorders) | 11 (25) | 7 (19)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 14 (41) | 15 (55)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (9) | 7 (22)
Blood disorder (Blood and lymphatic system disorders) | 4 (45) | 5 (12)
Bone pain (Musculoskeletal and connective tissue disorders) | 7 (20) | 7 (13)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 7 (10)
Chills (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 6 (12)
Confusion (Nervous system disorders) | 5 (6) | 6 (9)
Constipation (Gastrointestinal disorders) | 17 (32) | 20 (42)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (25) | 9 (17)
Dehydration (General disorders) | 6 (23) | 9 (13)
Depression (Nervous system disorders) | 9 (13) | 4 (9)
Diarrhea (Gastrointestinal disorders) | 17 (57) | 22 (33)
Dizziness (Nervous system disorders) | 8 (9) | 7 (18)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (8)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 4 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (24) | 10 (14)
ENT examination abnormal (Gastrointestinal disorders) | 10 (22) | 9 (14)
Edema, limbs (General disorders) | 1 (2) | 5 (6)
Fatigue (General disorders) | 25 (58) | 23 (57)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (9) | 9 (13)
Fever (General disorders) | 23 (56) | 18 (31)
Gingival infection (Infections and infestations) | 7 (9) | 3 (4)
Headache (General disorders) | 21 (48) | 17 (46)
Hemoglobin decreases (Blood and lymphatic system disorders) | 22 (141) | 28 (172)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 7 (12) | 2 (3)
Hyperbilirubinemia (Hepatobiliary disorders) | 4 (12) | 10 (25)
Hyperglycemia (Metabolism and nutrition disorders) | 14 (64) | 16 (55)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (23) | 9 (19)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (12) | 5 (15)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (25) | 14 (41)
Hypokalemia (Metabolism and nutrition disorders) | 11 (26) | 11 (42)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (8) | 4 (7)
Hyponatremia (Metabolism and nutrition disorders) | 9 (23) | 8 (14)
Hypotension (Cardiac disorders) | 13 (14) | 2 (2)
Infection (Infections and infestations) | 16 (44) | 23 (30)
Insomnia (General disorders) | 6 (13) | 13 (20)
Leukopenia (Blood and lymphatic system disorders) | 21 (142) | 23 (207)
Lymphatic disorder (General disorders) | 5 (10) | 6 (18)
Lymphopenia (Blood and lymphatic system disorders) | 10 (91) | 10 (142)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (12) | 3 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (9) | 11 (15)
Nausea (Gastrointestinal disorders) | 31 (85) | 24 (79)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 6 (7)
Neutropenia (Blood and lymphatic system disorders) | 28 (100) | 30 (133)
Oral pain (General disorders) | 4 (13) | 2 (2)
Pain (General disorders) | 6 (9) | 7 (16)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (8) | 5 (16)
Peripheral motor neuropathy (Nervous system disorders) | 2 (10) | 4 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 16 (57) | 20 (76)
Platelet count decreases (Blood and lymphatic system disorders) | 14 (58) | 20 (112)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (6) | 6 (10)
Rash desquamation (Skin and subcutaneous tissue disorders) | 13 (32) | 9 (14)
Sinus tachycardia (Cardiac disorders) | 7 (26) | 3 (6)
Skin disorder (Skin and subcutaneous tissue disorders) | 8 (18) | 5 (26)
Sweating (General disorders) | 11 (15) | 13 (29)
Taste alteration (Gastrointestinal disorders) | 6 (10) | 0 (0)
Thrombosis (Vascular disorders) | 3 (3) | 3 (5)
Urogenital disorder (Renal and urinary disorders) | 3 (4) | 3 (8)
Vomiting (Gastrointestinal disorders) | 20 (50) | 20 (42)
Weight loss (General disorders) | 7 (14) | 11 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less